CLINICAL TRIAL: NCT04497129
Title: Randomized Multicenter Comparative Trial Evaluating the Impact of the ROMTECH PortableConnect Rehabilitation Device on Time to Recovery and Comprehensive Rehabilitation Outcomes Post Unilateral Total Knee Arthroplasty (TKA)
Brief Title: ROMTECH PortableConnect Rehabilitation Device Usage Post Unilateral Total Knee Arthroplasty (TKA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ROM Technologies, INC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ROMTECH-0002
Record Dates: First submitted 2020-07-21; First posted 2020-08-04 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Knee Osteoarthritis; Knee Arthritis; Knee Pain Chronic; Knee Disease; Joint Pain; Osteo Arthritis Knee; Osteoarthritis, Knee
Keywords: ROMTech; PortableConnect; Osteoarthritis; Remote monitoring; Home Health Physical Therapy; Outpatient Physical Therapy; Rehabilitation; Physical Therapy
MeSH Terms: conditions — Osteoarthritis, Knee; Arthralgia; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- ROMTech PortableConnect (Experimental): Rehabilitation Using the ROMTech PortableConnect Device
  Interventions: Device: ROMTech PortableConnect
- Traditional Rehabilitation & Continuous Passive Motion Device (Active Comparator): Combination of OPPT and HHPT in conjunction with CPM device usage
  Interventions: Device: Traditional Rehabilitation and CPM Device

INTERVENTIONS:
Device: ROMTech PortableConnect — ROMTech PortableConnect (ROMTechPC) therapy will be completed four to five times per day for 6 minutes duration for 6 weeks. The intervention will be administered using the portable rehabilitation unit.
  Arms: ROMTech PortableConnect
Device: Traditional Rehabilitation and CPM Device — Continuous passive motion (CPM) with standard of care HHPT and OPPT rehabilitation program (CPM with SOC). Therapy with the CPM will be completed daily from day 0 through week 3 for a total of 6 to 8 hours per day. The HHPT and OPPT rehabilitation program will be a 6-week program based on SOC goals.
  Arms: Traditional Rehabilitation & Continuous Passive Motion Device

SUMMARY:
ROMTech is focused on transforming the healthcare market by delivering lower extremity rehabilitation systems that are effective, efficient for patient use, cost-effective, and provide better patient outcomes while simultaneously decreasing rehabilitation and overall recovery times.

DETAILED DESCRIPTION:
The patented technology of the ROMTech PortableConnect can improve the rehabilitation protocol for lower extremities in shorter time periods. The focus of this study is to compare the effectiveness of the ROMTech PortableConncect device only rehabilitation program following total knee arthroplasty to an active comparator group of continuous passive motion with a standard of care combination HHPT and OPPT rehabilitation program. The technology used to develop the ROMTech PortableConnect device has been reported in a pilot study to tend to be highly effective in decreasing the recovery time of patients post TKA, as discussed in the findings from the pilot study with the ROMTech Pro Cycle. The expedited recovery resulting from use of the ROMTech rehabilitation technology is noted to be contributed to the ability of the ROMTech technology to achieve a more rapid range of motion in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years of age at screening visit.
* Documentation of a definitive diagnosis of osteoarthritis of the knee requiring total knee arthroplasty.
* Scheduled or willing to schedule TKA procedure within the timelines consistent with the study enrollment period. This includes up to a 28-day screening window prior to the scheduled surgery.
* Willing to consent to outpatient, home-based physical therapy, CPM, or the ROMTech protocol
* Able to provide written informed consent.
* Willing and able to participate in and complete all study assessments, questionnaires, and procedure

Exclusion Criteria:

* Inability to provide informed consent.
* Inability to understand and complete study related assessments and procedures.
* Other scheduled surgical knee procedures in addition to the TKA.
* Presence of a condition or abnormality that in the opinion of the investigator would compromise the safety of the subject or the quality of the data.
* History of musculoskeletal or neurological disorders that limit physical function including but not limited to severe spine OA, contralateral leg issues limiting mobility, and other disorders as identified by the investigator
* Planned additional knee joint surgery within 3 months of the primary scheduled TKA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Range of Motion | Screening
  Knee Flexion and Extension
Range of Motion | Baseline
  Knee Flexion and Extension
Range of Motion | Week 1
  Knee Flexion and Extension
Range of Motion | Week 2
  Knee Flexion and Extension
Range of Motion | Week 3
  Knee Flexion and Extension
Range of Motion | Week 4
  Knee Flexion and Extension
Range of Motion | Week 5
  Knee Flexion and Extension
Range of Motion | Week 6
  Knee Flexion and Extension
Range of Motion | Week 7 (End of Treatment)
  Knee Flexion and Extension
Range of Motion | Week 9 (Follow-up)
  Knee Flexion and Extension

SECONDARY OUTCOMES:
Timed up and go (TUG) performance | Screening
  Assessment performed by study team
Timed up and go (TUG) performance | Week 4
  Assessment performed by study team
Timed up and go (TUG) performance | Week 7 (End of Treatment)
  Assessment performed by study team
Timed up and go (TUG) performance | Week 9 (Follow-UP)
  Assessment performed by study team
Knee pain as measured on a 10-point pain scale | Screening
  Patient reported outcome
Knee pain as measured on a 10-point pain scale | Baseline
  Patient reported outcome
Knee pain as measured on a 10-point pain scale | Week 1
  Patient reported outcome
Knee pain as measured on a 10-point pain scale | Week 2
  Patient reported outcome
Knee pain as measured on a 10-point pain scale | Week 3
  Patient reported outcome
Knee pain as measured on a 10-point pain scale | Week 4
  Patient reported outcome
Knee pain as measured on a 10-point pain scale | Week 5
  Patient reported outcome
Knee pain as measured on a 10-point pain scale | Week 6
  Patient reported outcome
Knee pain as measured on a 10-point pain scale | Week 7 (End of Treatment)
  Patient reported outcome
Knee pain as measured on a 10-point pain scale | Week 9 (Follow-up)
  Patient reported outcome
Knee swelling | Screening
  measured using a tape measure to obtain the circumference of the knee
Knee swelling | Baseline
  measured using a tape measure to obtain the circumference of the knee
Knee swelling | Week 1
  measured using a tape measure to obtain the circumference of the knee
Knee swelling | Week 2
  measured using a tape measure to obtain the circumference of the knee
Knee swelling | Week 3
  measured using a tape measure to obtain the circumference of the knee
Knee swelling | Week 4
  measured using a tape measure to obtain the circumference of the knee
Knee swelling | Week 5
  measured using a tape measure to obtain the circumference of the knee
Knee swelling | Week 6
  measured using a tape measure to obtain the circumference of the knee
Knee swelling | Week 7 (End of Treatment)
  measured using a tape measure to obtain the circumference of the knee
Knee swelling | Week 9 (Follow-up)
  measured using a tape measure to obtain the circumference of the knee
Lower extremity functionality as measured using the Lower Extremity Functionality Scale (LEFS) | Screening
  Patient reported outcome
Lower extremity functionality as measured using the Lower Extremity Functionality Scale (LEFS) | Baseline
  Patient reported outcome
Lower extremity functionality as measured using the Lower Extremity Functionality Scale (LEFS) | Week 1
  Patient reported outcome
Lower extremity functionality as measured using the Lower Extremity Functionality Scale (LEFS) | Week 2
  Patient reported outcome
Lower extremity functionality as measured using the Lower Extremity Functionality Scale (LEFS) | Week 3
  Patient reported outcome
Lower extremity functionality as measured using the Lower Extremity Functionality Scale (LEFS) | Week 4
  Patient reported outcome
Lower extremity functionality as measured using the Lower Extremity Functionality Scale (LEFS) | Week 5
  Patient reported outcome
Lower extremity functionality as measured using the Lower Extremity Functionality Scale (LEFS) | Week 6
  Patient reported outcome
Lower extremity functionality as measured using the Lower Extremity Functionality Scale (LEFS) | Week 7 (End of Treatment)
  Patient reported outcome
Lower extremity functionality as measured using the Lower Extremity Functionality Scale (LEFS) | Week 9 (Follow-up)
  Patient reported outcome
Ambulation using the 6 Minute Walk Test (6MWT) | Screening, Baseline
  Assessment performed by study team
Ambulation using the 6 Minute Walk Test (6MWT) | Baseline
  Assessment performed by study team
Ambulation using the 6 Minute Walk Test (6MWT) | Week 4
  Assessment performed by study team
Ambulation using the 6 Minute Walk Test (6MWT) | Week 7 (End of Treatment)
  Assessment performed by study team
Ambulation using the 6 Minute Walk Test (6MWT) | Week 9 (Follow-up)
  Assessment performed by study team
Days to ambulate without assistive devices and/or assistance | Screening
  Obtained via single response question
Days to ambulate without assistive devices and/or assistance | Baseline
  Obtained via single response question
Days to ambulate without assistive devices and/or assistance | Week 1
  Obtained via single response question
Days to ambulate without assistive devices and/or assistance | Week 2
  Obtained via single response question
Days to ambulate without assistive devices and/or assistance | Week 3
  Obtained via single response question
Days to ambulate without assistive devices and/or assistance | Week 4
  Obtained via single response question
Days to ambulate without assistive devices and/or assistance | Week 5
  Obtained via single response question
Days to ambulate without assistive devices and/or assistance | Week 6
  Obtained via single response question
Days to ambulate without assistive devices and/or assistance | Week 7 (End of Treatment)
  Obtained via single response question
Days to ambulate without assistive devices and/or assistance | Week 9 (Follow-up)
  Obtained via single response question
Days to return to activities of daily living | Screening
  Obtained via patient interview
Days to return to activities of daily living | Baseline
  Obtained via patient interview
Days to return to activities of daily living | Week 1
  Obtained via patient interview
Days to return to activities of daily living | Week 2
  Obtained via patient interview
Days to return to activities of daily living | Week 3
  Obtained via patient interview
Days to return to activities of daily living | Week 4
  Obtained via patient interview
Days to return to activities of daily living | Week 5
  Obtained via patient interview
Days to return to activities of daily living | Week 6
  Obtained via patient interview
Days to return to activities of daily living | Week 7 (End of Treatment)
  Obtained via patient interview
Days to return to activities of daily living | Week 9 (Follow-up)
  Obtained via patient interview
Opioid usage | Screening
  Compared to baseline opioid use by concomitant medication tracking at each visit
Opioid usage | Baseline
  Compared to baseline opioid use by concomitant medication tracking at each visit
Opioid usage | Week 1
  Compared to baseline opioid use by concomitant medication tracking at each visit
Opioid usage | Week 2
  Compared to baseline opioid use by concomitant medication tracking at each visit
Opioid usage | Week 3
  Compared to baseline opioid use by concomitant medication tracking at each visit
Opioid usage | Week 4
  Compared to baseline opioid use by concomitant medication tracking at each visit
Opioid usage | Week 5
  Compared to baseline opioid use by concomitant medication tracking at each visit
Opioid usage | Week 6
  Compared to baseline opioid use by concomitant medication tracking at each visit
Opioid usage | Week 7 (End of Treatment)
  Compared to baseline opioid use by concomitant medication tracking at each visit
Opioid usage | Week 9 (Follow-up)
  Compared to baseline opioid use by concomitant medication tracking at each visit
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Screening
  Patient reported outcome
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Baseline
  Patient reported outcome
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Week 1
  Patient reported outcome
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Week 2
  Patient reported outcome
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Week 3
  Patient reported outcome
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Week 4
  Patient reported outcome
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Week 5
  Patient reported outcome
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Week 6
  Patient reported outcome
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Week 7 (End of Treatment)
  Patient reported outcome
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Week 9 (Follow-up)
  Patient reported outcome
Oxford Knee Score (OKS) | Screening
  Patient reported outcome
Oxford Knee Score (OKS) | Baseline
  Patient reported outcome
Oxford Knee Score (OKS) | Week 1
  Patient reported outcome
Oxford Knee Score (OKS) | Week 2
  Patient reported outcome
Oxford Knee Score (OKS) | Week 3
  Patient reported outcome
Oxford Knee Score (OKS) | Week 4
  Patient reported outcome
Oxford Knee Score (OKS) | Week 5
  Patient reported outcome
Oxford Knee Score (OKS) | Week 6
  Patient reported outcome
Oxford Knee Score (OKS) | Week 7 (End of Treatment)
  Patient reported outcome
Oxford Knee Score (OKS) | Week 9 (Follow-up)
  Patient reported outcome

OTHER OUTCOMES:
Patient Satisfaction Questionnaire via 4-point scale | Week 1
  Patient Reported Outcome
Patient Satisfaction Questionnaire via 4-point scale | Week 2
  Patient Reported Outcome
Patient Satisfaction Questionnaire via 4-point scale | Week 3
  Patient Reported Outcome
Patient Satisfaction Questionnaire via 4-point scale | Week 4
  Patient Reported Outcome
Patient Satisfaction Questionnaire via 4-point scale | Week 5
  Patient Reported Outcome
Patient Satisfaction Questionnaire via 4-point scale | Week 6
  Patient Reported Outcome
Patient Satisfaction Questionnaire via 4-point scale | Week 7 (End of Treatment)
  Patient Reported Outcome
Patient Satisfaction Questionnaire via 4-point scale | Week 9 (Follow-up)
  Patient Reported Outcome
Manipulation under anesthesia | Baseline
  By patient questionnaires
Manipulation under anesthesia | Week 1
  By patient questionnaires
Manipulation under anesthesia | Week 2
  By patient questionnaires
Manipulation under anesthesia | Week 3
  By patient questionnaires
Manipulation under anesthesia | Week 4
  By patient questionnaires
Manipulation under anesthesia | Week 5
  By patient questionnaires
Manipulation under anesthesia | Week 6
  By patient questionnaires
Manipulation under anesthesia | Week 7 (End of Treatment)
  By patient questionnaires
Manipulation under anesthesia | Week 9 (Follow-up)
  By patient questionnaires
Total number of physical therapy sessions completed | Baseline
  A sum of all physical therapy sessions outpatient and home health visits
Total number of physical therapy sessions completed | Week 1
  A sum of all physical therapy sessions outpatient and home health visits
Total number of physical therapy sessions completed | Week 2
  A sum of all physical therapy sessions outpatient and home health visits
Total number of physical therapy sessions completed | Week 3
  A sum of all physical therapy sessions outpatient and home health visits
Total number of physical therapy sessions completed | Week 4
  A sum of all physical therapy sessions outpatient and home health visits
Total number of physical therapy sessions completed | Week 5
  A sum of all physical therapy sessions outpatient and home health visits
Total number of physical therapy sessions completed | Week 6
  A sum of all physical therapy sessions outpatient and home health visits
Total number of physical therapy sessions completed | Week 7 (End of Treatment)
  A sum of all physical therapy sessions outpatient and home health visits
Total number of physical therapy sessions completed | Week 9 (Follow-up)
  A sum of all physical therapy sessions outpatient and home health visits

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Nunley, MD, Study Director — ROM Tech
Locations (5):
- United States (5):
  - OrthoArizona, Gilbert, Arizona
  - Aventura Orthopaedics, Aventura, Florida
  - Orthopaedic Associates of West Florida, Clearwater, Florida
  - Institute of Orthopedic Research and Innovation, Coeur d'Alene, Idaho
  - OrthoSouth, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No